CLINICAL TRIAL: NCT03894150
Title: A Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of F0002-ADC in Chinese Patients With Refractory or Recurrent CD30+ Hematologic Malignancies.
Brief Title: A Study of F0002-ADC in Chinese Patients With Refractory or Recurrent CD30+ Hematologic Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F0002-01
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Refractory or Recurrent CD30+ Hematologic Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- F0002-ADC (Experimental)
  Interventions: Drug: F0002-ADC

INTERVENTIONS:
Drug: F0002-ADC — Every 21 days for 1 cycle, continue treatment until a maximum 16 cycles. Dose Escalating: 0.3 - 4.8 mg/kg

SUMMARY:
This is a Phase I dose escalation study designed to define the maximum tolerable dose(MDT), the safety profile, pharmacokinetic parameters, immunogenicity and anti-tumor activity of F0002-ADC in Chinese patients with relapsed/refractory CD30-positive hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* With relapsed/refractory CD30+ disease that histologically confirmed by central laboratory assessment and pathology review (Priority for cHL, ALCL and MF).
* Patients must have at least one site of measurable disease by conventional CT scan (defined by unidimensional lymph node lesion ≥ 15 mm or extranodal lesion ≥ 10 mm ), patients with MF, skin nodules can be measured by caliper to meet the criteria as measurable lesions, positive FDG uptake for cHL and ALCL.
* Patients must have the following required baseline laboratory data: Hb≥80g/L, NEUT≥1.5×109/L, PLT≥75×109/L, TBIL≤1.5 times ULN, ALT/AST≤2.5 times ULN, Cr≤1.25 times ULN or Ccr≥45 ml/min, INR≤1.5 times ULN, APTT≤1.5 times ULN.
* Patients must be at least 8 weeks apart from the previous autologous stem cell infusion therapy prior to the first dose.
* Patients must be at least 4 weeks apart from previous radiotherapy, chemotherapy, biologics, immunotherapy, and/or other research-based anticancer therapy prior to the first dose (with nitrogen mustard, melphalan, and nitrosourea for at least 6 weeks).
* Patients must have a life expectancy > 3 months.
* Voluntary consent form

Exclusion Criteria:

* Patients who have received an allogeneic stem cell transplant.
* Patients who have had previous treatment with any anti-CD30 antibody.
* Patients received antibody therapy 6 weeks or 5 plasma half-life before the first dose.
* Patients who are receiving other anti-tumor treatments.
* The toxicity of previous anti-tumor treatment has not recovered to grade 1 or below, except for grade 2 peripheral neurotoxicity and any level of alopecia.
* Other primary malignant tumors have been seen in the past 3 years (except for cervical cancer in situ or non-melanoma skin cancer or prostate cancer with specific prostate specific antigen).
* Participants with cardiovascular conditions specified in protocols.
* NYHA classification grading of cardiac function III/IV.
* Participants with brain or meningeal disease conditions specified in protocols.
* Patients with poor diabetes control,
* High-risk participants with a history of > grade 2 peripheral neuropathy or any active neurologic disease.
* Patients have psychiatric history.
* Patients with a history of liver fibrosis or cirrhosis and clinical signs and symptoms suggesting liver fibrosis or cirrhosis.
* Patients with previous interstitial pneumonia.
* Patients have active systemic viral, bacterial or fungal infection 4 weeks prior to the first dose
* HIV antibody positive / HBsAg positive / HCVAb positive.
* Patients who are allergic to recombinant proteins, murine proteins or to the drug excipients.
* Patients who are receiving a dose ≥ 20 mg/day of prednisone or glucocorticoid therapy.
* Female patients who are breastfeeding or pregnant.
* Patients with fertility who refuses to use contraception during the trial period and within 6 months after the end of the last dose.
* Other reasons that researchers believe are inappropriate to participate in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
MTD | Within 21 days after a single dose
  the maximum tolerable dose

SECONDARY OUTCOMES:
ORR | Once every 2 cycles and once every 4 cycles after 4 cycles (each cycle is 21 days), till tumor progression/death /3 years
  Objective response rate
DOR | Once every 2 cycles and once every 4 cycles after 4 cycles(each cycle is 21 days), till tumor progression/death /3 years
  Duration of Response
PFS | Once every 2 cycles and once every 4 cycles after 4 cycles(each cycle is 21 days), till tumor progression/death /3 years
  Progress Free Survival
Maximum Plasma Concentration [Cmax] | 1 months after last dose
  pharmacokinetic parameter
Area Under the Curve [AUC] | 1 months after last dose
  pharmacokinetic parameter
Tmax | 1 months after last dose
  pharmacokinetic parameter
Half-life Time [T1/2] | 1 months after last dose
  pharmacokinetic parameter
Clearance [CL] | 1 months after last dose
  pharmacokinetic parameter
Apparent Volume of Distribution [Vd] | 1 months after last dose
  pharmacokinetic parameter
Immunogenicity | 1 months after last dose
  Anti-F0002-ADC Antibodies
Incidence of adverse events | Till 1 month after last dose
Incidence of laboratory abnormalities | Till 1 month after last dose

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan